CLINICAL TRIAL: NCT00745693
Title: The Effects of Diesel Exhaust Inhalation on Vascular Function - the Role of Endothelin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Res08/A116
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2008-09

CONDITIONS: Coronary Disease
Keywords: Endothelin; Air pollution; Diesel exhaust; Vascular function; exposure
MeSH Terms: conditions — Coronary Disease | interventions — Endothelin-1; cyclo(Trp-Asp-Pro-Val-Leu); BQ 788

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 1 hour exposure to filtered air, followed by forearm venous occlusion plethysmography at 2 hours after the exposure and infusion of endothelin-1 (5pmol/min)
  Interventions: Drug: Endothelin-1
- 2 (Experimental): 1 hour exposure to filtered air, followed by forearm venous occlusion plethysmography at 2 hours after the exposure and infusion of endothelin receptor antagonists BQ-123 and BQ-788
  Interventions: Drug: BQ-123 and BQ-788
- 3 (Experimental): 1 hour exposure to dilute diesel exhaust (300mcg/m3), followed by forearm venous occlusion plethysmography at 2 hours after the exposure and infusion of endothelin-1 (5pmol/min)
  Interventions: Drug: Endothelin-1
- 4 (Experimental): 1 hour exposure to dilute diesel exhaust (300mcg/m3), followed by forearm venous occlusion plethysmography at 2 hours after the exposure and infusion of endothelin receptor antagonists BQ-123 and BQ-788
  Interventions: Drug: BQ-123 and BQ-788

INTERVENTIONS:
Drug: Endothelin-1 — Intra-arterial infusion of Endothelin-1 at 5pmol/min for 1 hour during venous occlusion plethysmography
  Other Names: ET-1; American Peptides - 88-1-10 (ET-1)
  Arms: 1; 3
Drug: BQ-123 and BQ-788 — 1 hour intra-arterial infusion of BQ-123 at 10nmol/min followed by co-infusion of BQ-788 at 1nmol/min for a further hour during forearm venous occlusion plethysmography
  Other Names: American Peptides - 88-2-10 (BQ-123); American Peptides - 88-2-55 (BQ-788)
  Arms: 2; 4

SUMMARY:
The purpose of this study is to identify the role of endothelin 1 (a natural vasoconstrictor) in the adverse vascular effects demonstrated after exposure to air pollution

DETAILED DESCRIPTION:
Air pollution is a major problem, and can be linked to around 5% of all deaths worldwide each year. There are strong associations between air pollution exposure and heart disease but we do not yet understand how these harmful effects are mediated. Understanding this mechanism is likely to have a major impact on the way we treat patients with heart disease and have the potential to shape future environmental health policy. The upregulation of Endothelin-1 provides a plausible mechanism for these harmful effects, and we plan to investigate this in more depth in the human forearm following exposure to diesel exhaust.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Use of regular medication
* Cigarette smoking
* Significant occupational exposure to air pollution
* Intercurrent illness

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow following infusion of endothelin-1 or the endothelin receptor antagonists BQ-123 & BQ-788 | 2 hours after exposure

SECONDARY OUTCOMES:
24 hour mean blood pressure (ambulatory monitoring) | 24 hours following the exposure
Systemic endothelin-1 and big endothelin-1 concentrations | At baseline, and immediately, 1, 2, 3, 4, 6 and 24 hours after exposure
Changes in arterial stiffness (pulse-wave velocity) | During and for the 1 hour after the exposure

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Langrish, MB BCh MRCP, Principal Investigator — University of Edinburgh; Anders Blomberg, MD, Study Director — Umeå University; Thomas Sandström, MD, Study Director — Umeå University; David E Newby, MD FRCP, Study Director — University of Edinburgh
Locations (1):
- Umeå University, Umeå, Västerbottens, Sweden

REFERENCES:
- [Background] Mills NL, Tornqvist H, Robinson SD, Gonzalez M, Darnley K, MacNee W, Boon NA, Donaldson K, Blomberg A, Sandstrom T, Newby DE. Diesel exhaust inhalation causes vascular dysfunction and impaired endogenous fibrinolysis. Circulation. 2005 Dec 20;112(25):3930-6. doi: 10.1161/CIRCULATIONAHA.105.588962. PMID 16365212
- [Background] Tornqvist H, Mills NL, Gonzalez M, Miller MR, Robinson SD, Megson IL, Macnee W, Donaldson K, Soderberg S, Newby DE, Sandstrom T, Blomberg A. Persistent endothelial dysfunction in humans after diesel exhaust inhalation. Am J Respir Crit Care Med. 2007 Aug 15;176(4):395-400. doi: 10.1164/rccm.200606-872OC. Epub 2007 Apr 19. PMID 17446340
- [Background] Calderon-Garciduenas L, Vincent R, Mora-Tiscareno A, Franco-Lira M, Henriquez-Roldan C, Barragan-Mejia G, Garrido-Garcia L, Camacho-Reyes L, Valencia-Salazar G, Paredes R, Romero L, Osnaya H, Villarreal-Calderon R, Torres-Jardon R, Hazucha MJ, Reed W. Elevated plasma endothelin-1 and pulmonary arterial pressure in children exposed to air pollution. Environ Health Perspect. 2007 Aug;115(8):1248-53. doi: 10.1289/ehp.9641. PMID 17687455
- [Background] Peretz A, Sullivan JH, Leotta DF, Trenga CA, Sands FN, Allen J, Carlsten C, Wilkinson CW, Gill EA, Kaufman JD. Diesel exhaust inhalation elicits acute vasoconstriction in vivo. Environ Health Perspect. 2008 Jul;116(7):937-42. doi: 10.1289/ehp.11027. PMID 18629317
- [Background] Vincent R, Kumarathasan P, Goegan P, Bjarnason SG, Guenette J, Berube D, Adamson IY, Desjardins S, Burnett RT, Miller FJ, Battistini B. Inhalation toxicology of urban ambient particulate matter: acute cardiovascular effects in rats. Res Rep Health Eff Inst. 2001 Oct;(104):5-54; discussion 55-62. PMID 11833973
- [Derived] Langrish JP, Lundback M, Mills NL, Johnston NR, Webb DJ, Sandstrom T, Blomberg A, Newby DE. Contribution of endothelin 1 to the vascular effects of diesel exhaust inhalation in humans. Hypertension. 2009 Oct;54(4):910-5. doi: 10.1161/HYPERTENSIONAHA.109.135947. Epub 2009 Aug 17. PMID 19687345